CLINICAL TRIAL: NCT02964884
Title: Neurobiology and Treatment of Reading Disability in NF1
Brief Title: Interventions for Reading Disabilities in NF1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laura Cutting, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 161159; 1R01HD089474-01 (NIH)
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Neurofibromatosis Type 1; Learning Disability; Reading Disability; NF1
Keywords: Neurofibromatosis Type 1; Learning Disability; Reading Disability; NF1
MeSH Terms: conditions — Neurofibromatosis 1; Learning Disabilities; Dyslexia | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NF1: Lovastatin + reading tutoring (Active Comparator): Participants (NF-1 patients) will receive 20mg of Lovastatin per day for the first two weeks, the dose will be escalated 40 mg for the remaining 11 weeks.
  And one week of intensive, one-on-one reading tutoring intervention
  Interventions: Drug: Lovastatin; Behavioral: reading tutoring intervention
- NF1: Placebo + reading tutoring (Placebo Comparator): Participants (NF-1 patients) will receive placebo daily And one week of intensive, one-on-one reading tutoring intervention
  Interventions: Behavioral: reading tutoring intervention; Drug: Placebo Oral Tablet
- RD: Reading tutoring (Placebo Comparator): Participants (RD-only participants) will receive one week of intensive, one-on-one reading tutoring intervention
  Interventions: Behavioral: reading tutoring intervention
- RD: Other Academic (sham) tutoring (Sham Comparator): Participants (RD-only participants) will receive one week of intensive, one-on-one tutoring intervention with an academic focus other than reading.
  These participants will have the opportunity to receive reading tutoring upon finishing study participation.
  Interventions: Behavioral: Other Academic "sham" tutoring

INTERVENTIONS:
Drug: Lovastatin — Those in the Lovastatin group will receive 20mg of Lovastatin per day for the first two weeks and 40mg of Lovastatin per day starting at week 3 through week 11.
  Arms: NF1: Lovastatin + reading tutoring
Behavioral: reading tutoring intervention — After the initial 12 weeks of Lovastatin or placebo, children will return for one week of intensive, one-on-one tutoring intervention (either reading or sham; Visit 2)
  Arms: NF1: Lovastatin + reading tutoring; NF1: Placebo + reading tutoring; RD: Reading tutoring
Drug: Placebo Oral Tablet — Those in the placebo group will receive a tablet daily
  Arms: NF1: Placebo + reading tutoring
Behavioral: Other Academic "sham" tutoring — No reading (sham) tutoring. Children will receive intensive tutoring on a subject other than reading.
  Arms: RD: Other Academic (sham) tutoring

SUMMARY:
Neurofibromatosis Type 1 (NF1) is a common genetic disorder that is associated with a four times greater risk of learning disabilities, including reading disabilities, and a deficiency of neurofibromin - a protein important in a signaling pathway that regulates learning and memory. Our previous work (NS49096) demonstrated that school-age children with NF+RD can respond to standard phonologically-based reading tutoring originally developed to treat reading disability in the general population. Combining our work with that by other researchers suggesting that a medication (Lovastatin) may counteract the effects of the deficient neurofibromin, and possibly ameliorate learning disabilities in NF1, the investigator propose to examine the synergistic effects of medication plus reading tutoring.

DETAILED DESCRIPTION:
Neurofibromitosis Type 1 (NF1) is a common autosomal dominant neurocutaneous syndrome. The most common concern of NF1 is learning disabilities (LDs). Approximately half of children with NF1 have LDs, the most common of which are reading disabilities (RDs).The purpose of this research is to gain a deeper understanding of the characteristics and treatment of RDs in NF1.

The Investigator will evaluate four different groups (see list below) to determine if there are differential outcomes in these groups of children with NF+RD. The first two groups will consist of NF1 patients, and the second two groups will consist of participants with RDs but without NF1.

1. Reading tutoring program and a medication called Lovastatin (NF1 patients)
2. Reading tutoring program and no Lovastatin (placebo) (NF1 patients)
3. Reading tutoring program (RD participants)
4. Other Academic "Sham" tutoring (eligible to receive reading tutoring after study participation is complete) (RD participants)

ELIGIBILITY:
Inclusion Criteria:

This study will be open to all English speakers who meet eligibility criteria regardless of race, gender, minority or socioeconomic status. Inclusion criteria to be met are listed below:

1. Individuals ages 8-20 (all participants)
2. Documented NF-1 (NF patients only)
3. If female, participant is post-menarche (NF patients only)
4. If male, participant has reached Tanner Stage 2 (NF patients only)
5. Participant able to swallow capsule (NF patients only, may be confirmed via swallowability test, described below)
6. Participant's English is sufficient for school (all participants)
7. Participant must either answer "yes" to question A, or answer "yes" to at least 2 items for questions B-D listed below:

A. Has your child ever been diagnosed with a reading disability? B. Did your child have trouble learning how to "sound out" words? C. Have you (parent) ever been concerned about your child's reading ability? D. Did the school or teacher ever express any concerns about your child's reading ability? Swallowability Assessment: We may ask patients to perform a capsule swallowability assessment prior to enrollment. We will ask subjects to attempt to swallow an empty capsule, matching the same size of the Lovastatin 20mg and 40mg capsules to be used in the study, to confirm swallowability. Patients will be provided with up to 2 capsules as needed to successfully perform the swallowability assessment. If the patient is unable to swallow the capsule, enrollment in the study may deferred or declined.

A child will be excluded if he/she meets any of the following criteria, which will be determined by initial telephone screening as well as review of medical/developmental history prior to and during testing:

1. Child 7 years of age or less;
2. known uncorrectable visual impairment;
3. documented hearing impairment greater than or equal to a 25 dB loss;
4. medical contraindication to MRI procedures (e.g., metal devices);
5. any psychiatric, behavioral, or developmental disorder that would preclude active participation in in-depth tutoring sessions
6. Pregnant at time of screening.
7. Known conditions which are contraindicated to Lovastatin

   1. Hypersensitivity to the medication
   2. Uncontrolled Epilepsy
   3. Metabolic Syndrome X, High Blood Sugar,
   4. Muscle Damage Due to Autoimmunity
   5. Stroke caused by Bleeding in the Brain, Loss of Memory,
   6. Severely Low Blood Pressure
   7. Liver Problems including Abnormal Liver Function Tests
   8. Severe Renal Impairment,
   9. Serious Muscle Damage that may Lead to Kidney Failure,
   10. Recent Operation or significant Injury
   11. Muscle Pain or Tenderness with Increase Creatinine Kinase,
   12. Habit of Drinking Too Much Alcohol
   13. Pregnant or lactating. - Lovastatin is contraindicated during pregnancy and in nursing mothers because it decreases synthesis of cholesterol and other products of the cholesterol biosynthesis pathway that are essential components for fetal development.

Children who meet criteria for ADHD, Oppositional Defiant Disorder, adjustment disorder, and/or mild depression will be eligible as long as they are not taking psychotropic medications, with the exception of stimulant medication for ADHD.

For pilot participants only:

Criteria for inclusion/exclusion for pilot participants is outlined below. Children who meet criteria for ADHD, Oppositional Defiant Disorder, adjustment disorder, and/or mild depression will be eligible as long as they are not taking psychotropic medications, with the exception of stimulant medication for ADHD.

1. Children ages 8-17
2. Participant is a native English speaker
3. Participant must either answer "yes" to question A, or answer "yes" to at least 2 items for questions 2-4 listed below:

A. Has your child ever been diagnosed with a reading disability? B. Did your child have trouble learning how to "sound out" words? C. Have you (parent) ever been concerned about your child's reading ability? D. Did the school or teacher ever express any concerns about your child's reading ability?

A child will be excluded if he/she meets any of the following criteria, which will be determined by initial telephone screening as well as review of medical/developmental history prior to and during testing:

1. Children 7 years of age or younger
2. previous diagnosis of Intellectual Disability;
3. known uncorrectable visual impairment;
4. documented hearing impairment greater than or equal to a 25 dB loss;
5. medical contraindication to MRI procedures (e.g., metal devices);
6. known IQ below 70;
7. a pervasive developmental disorder; and
8. any known neurologic pathology, including epilepsy, spina bifida, cerebral palsy, traumatic brain injury, optic gliomas, and brain tumors (other than UBOs).
9. Comorbid severe psychiatric disorders will also be excluded.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Woodcock Johnson Tests of Achievement IV | 24 weeks
  WJ-IV (Forms A and B) Letter Word Identification, Word Attack, and Passage Comprehension subtests will be administered in order to assess word recognition accuracy, decoding accuracy, and comprehension.
Woodcock Reading Mastery Test-III | 24 weeks
  (WRMT-III; Forms A and B); Word Identification, Word Attack, and Passage Comprehension will be administered to assess word recognition accuracy, decoding accuracy, and comprehension. The WRMT-III and WJ-III correlate at .87, and at the item level show similar characteristics (e.g., containing 31% and 34% multisyllabic words, respectively).
Test of Word Reading Efficiency-2 | 24 weeks
  (TOWRE-2; Forms A, B, C, D) Sight Word Efficiency and Pseudoword Decoding will be used to assess real and pseudoword reading speed.
Experimental Word and Pseudoword Lists | 24 weeks
  At each visit, 2 word and 2 pseudoword lists (20 words each) will be administered. Word lists are matched on relevant characteristics (e.g., frequency, bigram frequency). Real word lists have already been developed and tested, and show high inter-correlations (r =.87-.97).
Test of Silent Contextual Reading Fluency-2 | 24 weeks
  (TOSCRF-2; 91; Forms A, B, C, D). This test requires identifying as many words as possible in 3 min within a sentential context.
Comprehensive Test of Phonological Processing-2 | 24 weeks
  CTOPP-2 core subtests will be used to assess phonological processing, a known predictor of decoding and word recognition.
Delis Kaplan Executive Function System | 24 weeks
  Sorting from the D-KEFS will be used to assess higher-level planning and shifting abilities.
Visuospatial Learning and Memory, Morris Water Maze | 24 weeks
  The child "hops" from square to square in the grid, repeated from various starting points. After landing on the target square, a fun goal pops up. The number of "hops" to reach the goal is measured. A control probe trial is given in which there is no goal.
Visuospatial Learning and Memory, Judgment of Line Orientation | 24 weeks
  (JLO, Forms J and H)98 requires the judgment of spatial relationships between two lines compared to a reference of a protractor-like half-circle of 11 lines. The Investigator will create 4 forms from the two already existing by splitting each test in half by selecting every other item, a method used by others (Leach et al., 2003). This will allow us to generate 4 different versions of the JLO.
Clinical Evaluation of Language Fundamentals-Fifth Edition | 24 weeks
  CELF-5 will be used to assess aspects of oral language (e.g., syntax, semantics, & working memory).

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Cutting, PhD, Principal Investigator — Vanderbilt University Medical Center; Sheryl L. Rimrodt-Frierson, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No